CLINICAL TRIAL: NCT05281120
Title: Low-level Mechanical Vibration, Bone Density, Bone Resorption and Muscular Strength in Ambulant Children Affected by Duchenne Muscular Dystrophy
Brief Title: Effects of Low-level Mechanical Vibration on Bone Density in Ambulant Children Affected by Duchenne Muscular Dystrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 02C701
Record Dates: First submitted 2022-02-18; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Osteoporosis; Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; children; low bone mass; osteoporosis; low-level mechanical vibration; bone turnover markers
MeSH Terms: conditions — Osteoporosis; Muscular Dystrophy, Duchenne

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (2):
- mechanical intervention group (Active Comparator): 20 subjects participated to the study (1 year double-blind, randomized, placebo controlled, parallel group study) and 10 subjects were randomized to this arm.
  Intervention: to stand on the active platform (inducing vertical, sinusoidal acceleration) for 10 minutes each day for 12 months.
  Interventions: Device: Low-level mechanical vibrations WITH vertical sinusoidal acceleration
- mechanical placebo group (Placebo Comparator): 20 subjects participated to the study (1 year double-blind, randomized, placebo controlled, parallel group study) and 10 subjects were randomized to this arm.
  Intervention: to stand on the placebo platform (not inducing vertical, sinusoidal acceleration) for 10 minutes each day for 12 months.
  Interventions: Device: Low-level mechanical vibrations WITHOUT vertical sinusoidal acceleration

INTERVENTIONS:
Device: Low-level mechanical vibrations WITH vertical sinusoidal acceleration — Small platform designed to induce vertical, sinusoidal acceleration.
  Arms: mechanical intervention group
Device: Low-level mechanical vibrations WITHOUT vertical sinusoidal acceleration — Small platform designed to NOT induce vertical, sinusoidal acceleration
  Arms: mechanical placebo group

SUMMARY:
Duchenne muscular dystrophy (DMD) is a X-linked recessive disorder due to a mutation of the dystrophin gene (Xp21). Dystrophin is a sarcolemmal protein of skeletal and cardiac muscle, and its absence causes progressive muscle degeneration and substitution with fat and connective tissue. The progressive muscle degeneration leads to loss of autonomous walking before the age of 15 years and death for cardiac and/or respiratory failure. There are no specific treatment for DMD, and the standard of care is now based on long-term corticosteroid (CS) use. The studies on bone mass in DMD are very few, but they agree in reporting the presence of a reduced bone mass and an increased rate of fractures probably due to long-term steroid therapy and disuse-osteopenia. The aim of this study, involving 20 ambulant DMD boys (age 7-10 years) has been the evaluation of the effects of low-level mechanical vibrations on bone in a group of ambulant DMD children for 1 year, with RDA-adjusted dietary calcium intake and 25OH vitamin D supplementation.

DETAILED DESCRIPTION:
All children were instructed to have a daily intake of calcium equal to the 100% of the RDA and were supplemented with calcifediol (0.7 mcg/kg/die).

The 20 boys were randomly assigned to two groups:

group 1 (mechanical intervention group) = a mechanical device (a small platform designed to induce vertical, sinusoidal acceleration) was installed in the home of each boy of group 1.

group 2 (placebo control group) = a placebo device was installed in the home of each boy of group 2

All boys were instructed to stand on the platform for 10 minutes each day for 12 months.

Compliance was followed and stimulated through weekly telephone contacts with parents and children.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DMD
* Ability to stand up and walk (some balance assistance allowed, but full weight-bearing necessary)
* All the children must already be on glucocorticoid therapy for at least 6 months before the start of the study.

Exclusion Criteria:

* Presence of other diseases interfering with bone density and bone turnover
* The inability to regularly use the vibratory platform.

Ages: 7 Years to 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2006-11; Primary Completion 2007-05 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Change in bone mineral density at lumbar spine. | baseline and 12th month
  Bone mineral density evaluated by DXA. Bone mineral apparent density calculated to correct for bone size (growing subjects). Z-score calculated.
  Measurements: baseline and 12 months.

SECONDARY OUTCOMES:
Calcium | baseline and 12th month
  changes in serum calcium (mg/dL)
Phosphate | baseline and 12th month
  changes in serum phosphate (mg/dL)
Magnesium | baseline and 12th month
  changes in serum magnesium (mg/dL)
Creatinine | baseline and 12th month
  changes in serum creatinine (mg/dL)
Bone Alkaline Phosphatase | baseline and 12th month
  changes in serum bone alkaline phosphatase (µg/L)
Osteocalcin | baseline and 12th month
  changes in serum osteocalcin (µg/L)
Parathyroid Hormone | baseline and 12th month
  changes in serum parathyroid hormone (ng/L)
25-OH vitamin D | baseline and 12th month
  changes in serum 25-OH vitamin D (µg/L)
1,25(OH)2 vitamin D | baseline and 12th month
  changes in serum 1,25(OH)2 vitamin D (ng/L)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Luisa Bianchi, Principal Investigator — Istituto Auxologico Italiano

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khan MA. Corticosteroid therapy in Duchenne muscular dystrophy. J Neurol Sci. 1993 Dec 1;120(1):8-14. doi: 10.1016/0022-510x(93)90017-s. PMID 8289083
- [Background] Mendell JR, Moxley RT, Griggs RC, Brooke MH, Fenichel GM, Miller JP, King W, Signore L, Pandya S, Florence J, et al. Randomized, double-blind six-month trial of prednisone in Duchenne's muscular dystrophy. N Engl J Med. 1989 Jun 15;320(24):1592-7. doi: 10.1056/NEJM198906153202405. PMID 2657428
- [Background] Bonifati MD, Ruzza G, Bonometto P, Berardinelli A, Gorni K, Orcesi S, Lanzi G, Angelini C. A multicenter, double-blind, randomized trial of deflazacort versus prednisone in Duchenne muscular dystrophy. Muscle Nerve. 2000 Sep;23(9):1344-7. doi: 10.1002/1097-4598(200009)23:93.0.co;2-f. PMID 10951436
- [Background] Biggar WD, Gingras M, Fehlings DL, Harris VA, Steele CA. Deflazacort treatment of Duchenne muscular dystrophy. J Pediatr. 2001 Jan;138(1):45-50. doi: 10.1067/mpd.2001.109601. PMID 11148511
- [Background] Consensus development conference: diagnosis, prophylaxis, and treatment of osteoporosis. Am J Med. 1993 Jun;94(6):646-50. doi: 10.1016/0002-9343(93)90218-e. No abstract available. PMID 8506892
- [Background] Baylink DJ. Glucocorticoid-induced osteoporosis. N Engl J Med. 1983 Aug 4;309(5):306-8. doi: 10.1056/NEJM198308043090509. No abstract available. PMID 6866054
- [Background] Chesney RW, Mazess RB, Rose P, Jax DK. Effect of prednisone on growth and bone mineral content in childhood glomerular disease. Am J Dis Child. 1978 Aug;132(8):768-72. doi: 10.1001/archpedi.1978.02120330040010. PMID 685891
- [Background] Jones G, Ponsonby AL, Smith BJ, Carmichael A. Asthma, inhaled corticosteroid use, and bone mass in prepubertal children. J Asthma. 2000;37(7):603-11. doi: 10.3109/02770900009090816. PMID 11059528
- [Background] Naganathan V, Jones G, Nash P, Nicholson G, Eisman J, Sambrook PN. Vertebral fracture risk with long-term corticosteroid therapy: prevalence and relation to age, bone density, and corticosteroid use. Arch Intern Med. 2000 Oct 23;160(19):2917-22. doi: 10.1001/archinte.160.19.2917. PMID 11041898
- [Background] Whalen RT, Carter DR, Steele CR. Influence of physical activity on the regulation of bone density. J Biomech. 1988;21(10):825-37. doi: 10.1016/0021-9290(88)90015-2. PMID 3225269
- [Background] Slemenda CW, Miller JZ, Hui SL, Reister TK, Johnston CC Jr. Role of physical activity in the development of skeletal mass in children. J Bone Miner Res. 1991 Nov;6(11):1227-33. doi: 10.1002/jbmr.5650061113. PMID 1805545
- [Background] Slemenda CW, Reister TK, Hui SL, Miller JZ, Christian JC, Johnston CC Jr. Influences on skeletal mineralization in children and adolescents: evidence for varying effects of sexual maturation and physical activity. J Pediatr. 1994 Aug;125(2):201-7. doi: 10.1016/s0022-3476(94)70193-8. PMID 8040762
- [Background] Courteix D, Lespessailles E, Peres SL, Obert P, Germain P, Benhamou CL. Effect of physical training on bone mineral density in prepubertal girls: a comparative study between impact-loading and non-impact-loading sports. Osteoporos Int. 1998;8(2):152-8. doi: 10.1007/BF02672512. PMID 9666939
- [Background] Palmieri GM, Bertorini TE, Griffin JW, Igarashi M, Karas JG. Assessment of whole body composition with dual energy x-ray absorptiometry in Duchenne muscular dystrophy: correlation of lean body mass with muscle function. Muscle Nerve. 1996 Jun;19(6):777-9. doi: 10.1002/(SICI)1097-4598(199606)19:63.0.CO;2-I. No abstract available. PMID 8609931
- [Background] Larson CM, Henderson RC. Bone mineral density and fractures in boys with Duchenne muscular dystrophy. J Pediatr Orthop. 2000 Jan-Feb;20(1):71-4. PMID 10641693
- [Background] Aparicio LF, Jurkovic M, DeLullo J. Decreased bone density in ambulatory patients with duchenne muscular dystrophy. J Pediatr Orthop. 2002 Mar-Apr;22(2):179-81. PMID 11856925
- [Background] McDonald DG, Kinali M, Gallagher AC, Mercuri E, Muntoni F, Roper H, Jardine P, Jones DH, Pike MG. Fracture prevalence in Duchenne muscular dystrophy. Dev Med Child Neurol. 2002 Oct;44(10):695-8. doi: 10.1017/s0012162201002778. PMID 12418795
- [Background] Welten DC, Kemper HC, Post GB, Van Mechelen W, Twisk J, Lips P, Teule GJ. Weight-bearing activity during youth is a more important factor for peak bone mass than calcium intake. J Bone Miner Res. 1994 Jul;9(7):1089-96. doi: 10.1002/jbmr.5650090717. PMID 7942156
- [Background] Vestergaard P, Glerup H, Steffensen BF, Rejnmark L, Rahbek J, Moseklide L. Fracture risk in patients with muscular dystrophy and spinal muscular atrophy. J Rehabil Med. 2001 Jul;33(4):150-5. PMID 11506212
- [Background] Talim B, Malaguti C, Gnudi S, Politano L, Merlini L. Vertebral compression in Duchenne muscular dystrophy following deflazacort. Neuromuscul Disord. 2002 Mar;12(3):294-5. doi: 10.1016/s0960-8966(01)00307-8. No abstract available. PMID 11801403
- [Background] Bianchi ML, Mazzanti A, Galbiati E, Saraifoger S, Dubini A, Cornelio F, Morandi L. Bone mineral density and bone metabolism in Duchenne muscular dystrophy. Osteoporos Int. 2003 Sep;14(9):761-7. doi: 10.1007/s00198-003-1443-y. Epub 2003 Jul 29. PMID 12897980
- [Background] Merlini L, Mazzone ES, Solari A, Morandi L. Reliability of hand-held dynamometry in spinal muscular atrophy. Muscle Nerve. 2002 Jul;26(1):64-70. doi: 10.1002/mus.10166. PMID 12115950
- [Background] Xie L, Jacobson JM, Choi ES, Busa B, Donahue LR, Miller LM, Rubin CT, Judex S. Low-level mechanical vibrations can influence bone resorption and bone formation in the growing skeleton. Bone. 2006 Nov;39(5):1059-1066. doi: 10.1016/j.bone.2006.05.012. Epub 2006 Jul 7. PMID 16824816
- [Background] Gilsanz V, Wren TA, Sanchez M, Dorey F, Judex S, Rubin C. Low-level, high-frequency mechanical signals enhance musculoskeletal development of young women with low BMD. J Bone Miner Res. 2006 Sep;21(9):1464-74. doi: 10.1359/jbmr.060612. PMID 16939405
- [Background] Ward K, Alsop C, Caulton J, Rubin C, Adams J, Mughal Z. Low magnitude mechanical loading is osteogenic in children with disabling conditions. J Bone Miner Res. 2004 Mar;19(3):360-9. doi: 10.1359/JBMR.040129. Epub 2004 Jan 27. PMID 15040823